CLINICAL TRIAL: NCT00970606
Title: Randomized, Placebo Controlled Trial of the Effectiveness of Statins for Preventing Mortality Following ICU Admission for Influenza Complications
Brief Title: STIP: Statin Trial for Influenza Patients
Acronym: STIP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit participants since H1N1 epidemic resolved.
Sponsor: Gordon Bernard (Other)
Responsible Party: Sponsor-Investigator, Gordon Bernard, Professor of Medicine, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STIP
Record Dates: First submitted 2009-08-31; First posted 2009-09-02 (Estimated); Results first posted 2013-04-24 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2013-06

CONDITIONS: Acute Respiratory Distress Syndrome; Influenza; H1N1 Influenza
Keywords: ARDS; H1N1; Influenza; Statin
MeSH Terms: conditions — Respiratory Distress Syndrome; Influenza, Human; Orthomyxoviridae Infections | interventions — Rosuvastatin Calcium; Sugars

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo tablet (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Rosuvastatin (crestor) (Experimental): Experimental arm
  Interventions: Drug: Rosuvastatin (crestor)

INTERVENTIONS:
Drug: Rosuvastatin (crestor) — 20 mg tablets once daily x max 28 days or for an additional 3 days following ICU discharge
  Other Names: Crestor
  Arms: Rosuvastatin (crestor)
Drug: Placebo — Placebo tablet identical to active therapy. 1 tablet per day
  Other Names: Placebo, sugar pill
  Arms: Placebo tablet

SUMMARY:
To assess the efficacy and safety of oral rosuvastatin in patients with suspected or confirmed influenza who require intensive care unit (ICU) admission due to respiratory distress.

DETAILED DESCRIPTION:
Hypothesis: Rosuvastatin therapy will improve mortality and reduce the need for mechanical ventilation in patients experiencing respiratory distress as a complication of influenza.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with suspected or confirmed influenza (Appendix A)
2. Requirement for ICU (or ICU step-down) admission due to respiratory distress defined as:

   * SaO2/FiO2 < 315 or PaO2/FiO2 < 300
   * Multiply by PB/760 (when altitude exceeds 51000 ft)
   * For FiO2 for non-intubated patients see Appendix B

Participants must receive the first dose of study drug within 48 hours following ICU admission for confirmed or suspected influenza or be excluded from participation in the study.

Exclusion Criteria:

1. No consent/inability to obtain consent
2. Age less than 13 years
3. Weight less than 40 kg
4. Unable to receive or unlikely to absorb enteral study drug (e.g. patients with partial or complete mechanical bowel obstruction, intestinal ischemia, infarction, and short bowel syndrome)
5. Allergy or intolerance to statins*
6. Pregnancy or breast feeding
7. Receiving niacin, fenofibrate, cyclosporine, gemfibrozil, or any antiviral protease inhibitor including but not limited to lopinavir and ritonavir.
8. Existing clinically significant myositis or myopathy or has a measured CK greater than 5,000 U/L
9. Requiring statin for underlying disease as determined by the patients attending physician team**.
10. Severe chronic liver disease (Child-Pugh Score 11-15)
11. Previous myocardial infarction or thrombotic stroke within the past 6 months 11.12. Any significant funding in the patient's medical history or physical or psychiatric exam prior to randomization that, in the opinion of the investigator, would affect patient safety or compliance or ability to deliver the study drug according to protocol

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon R Bernard, M.D., Principal Investigator — Vanderbilt University
Locations (21):
- United States (21):
  - University of Arkansas, Little Rock, Alaska
  - Maricopa Integrated Health System, Phoenix, Arizona
  - Stanford, Stanford, California
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins Hospital, Baltiomore, Maryland
  - Boston University, Boston, Massachusetts
  - Baystate Medical Center, Springfiled, Massachusetts
  - Columbia University, New York, New York
  - Mt Sinai, New York, New York
  - Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - Metro Health, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Oregon, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Erlanger, Chattanooga, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas, San Antonio, Texas
  - Intermountain, Murray, Utah
  - University of Virginia, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study terminated due to lack of recruitment due to earlier than anticipated end to H1N1 flu season
Groups:
- Placebo Tablet: Placebo
  Placebo : Placebo tablet identical to active therapy. 1 tablet per day
- Rosuvastatin (Crestor): Experimental arm
  Rosuvastatin (crestor) : 20 mg tablets once daily x max 28 days or for an additional 3 days following ICU discharge
Period: Overall Study
Arm/Group | Placebo Tablet | Rosuvastatin (Crestor)
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Tablet | Rosuvastatin (Crestor) | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.03 (12.89) | 39.88 (5.32) | 41.68 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Hospital Mortality to Day 28 or if Mortality is Not Different Between Groups, Time to Achieve Resolution of Respiratory Failure (e.g., Time to Unassisted Breathing in Survivors (Including Patient's Never Requiring Mechanical Ventilation).
Description: No outcome analyses were run as the sample size was not of sufficient size for a comparison with only 7 of >2000 participants planned/anticipated actually enrolled.
Time Frame: 28 days
Population: Only 7 participants were enrolled in this study designed for >2000. No formal anlaysis of outcomes was performed as tne n was too small to show any differences
Arm/Group | Placebo Tablet | Rosuvastatin (Crestor)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Placebo Tablet | Rosuvastatin (Crestor)
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 1/4 | 0/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Tablet (N=4) | Rosuvastatin (Crestor) (N=3)
Increased liver enzymes-AST/ALT (Hepatobiliary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Only able to enroll only 7 participants of >2000 planned/anticipated, leading to early termination of the study and therefore unable to perform statistical analysis with such a small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No